CLINICAL TRIAL: NCT04111978
Title: MAintenance Therapy With Aromatase Inhibitor in Epithelial Ovarian Cancer: a Randomized Double-blinded Placebo-controlled Multi-centre Phase III Trial (ENGOT-ov54/Swiss-GO-2/MATAO), Including LOGOS (Low Grade Ovarian Cancer Sub-study).
Brief Title: MAintenance Therapy With Aromatase Inhibitor in Epithelial Ovarian Cancer (MATAO)
Acronym: MATAO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss GO Trial Group (Network)
Collaborators: AGO Study Group (Other); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); Reliable Cancer Therapies (Industry); Krebsliga Schweiz (Unknown); Stiftung Guido Feger (Unknown); Hoffmann-La Roche (Industry); Helsana AG (Unknown); Novartis Pharmaceuticals (Industry); Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENGOT-ov54/Swiss-GO-2/MATAO; 2024-511219-78-00 (EU CTIS Number); 2019-002264-27 (EudraCT Number); ENGOT-ov54 (Other: European Network for Gynaecological Oncological Trial Groups); Swiss-GO-2 (Other: Swiss Network for Gynaecological Oncological Studies); AGO-OVAR 26 (Other: AGO Deutschland); AGO 65 (Other: AGO Austria)
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Neoplasm Epithelial; Fallopian Tube Neoplasms; Peritoneal Neoplasms; High-grade Serous Ovarian Carcinoma (HGSOC); Low-grade Serous Ovarian Carcinoma (LGSOC); Ovarian Endometrioid Carcinoma
Keywords: maintenance therapy; aromatase inhibitor; primary ovarian cancer; estrogen-receptor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (aromatase inhibitor) (Experimental): Letrozole, 2.5 mg Femara tablet, administered once daily for 5 years or until symptoms of toxicity or progression of underlying disease
  Interventions: Drug: Letrozole 2.5mg
- Placebo (Placebo Comparator): Placebo tablet of Femara (without aromatase inhibitor), 0 mg Femara tablet, administered once daily for 5 years or progression of underlying disease
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Letrozole 2.5mg — Aromatase inhibitor
  Other Names: Femara
  Arms: Letrozole (aromatase inhibitor)
Other: Placebo — Placebo tablet of Femara
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of addition of letrozole to the standard maintenance therapy in subjects following a primary diagnosis of Estrogen-receptor (ER) positive high and low grade epithelial ovarian cancer (including fallopian tube and primary peritoneal cancer) and subsequent primary treatment surgery and chemotherapy. Half of the participants will receive to the standard maintenance treatment, letrozole, whilst the other half receives placebo.

The study's primary hypothesis is that the treatment with letrozole increases progression free survival in comparison to the maintenance standard treatment (superiority trial).

DETAILED DESCRIPTION:
Femara (letrozole) is an extensively investigated, marketed aromatase inhibitor (AI) widely used as treatment in the maintenance phase of estrogen-receptor (ER) positive breast cancer, as it inhibit the synthesis of estrogens. Estrogen is a well known driver of cancer growth in ER-positive tumors and a high percentage of the epithelial ovarian cancers express ER as well. Of which low grade ovarian cancers demonstrates the highest level of expression, supporting our strategy of a sub-group analysis (LOGOS). Therefore, letrozole in this study be investigated prospectively and evaluated as maintenance therapy after standard surgical and chemotherapy treatment in comparison to placebo (which is the current standard maintenance treatment) in subjects with primary, ER-positive low or high grade serous or endometrioid epithelial ovarian cancer (including fallopian tube and primary peritoneal cancer) of FIGO Stage II-IV, whose cancer has not progressed by the end of the platinum-based chemotherapy.

The objectives are to evaluate the letrozole maintenance treatment compared to placebo in terms of

* progression-free survival (PFS; primary endpoint)
* overall survival (OS)
* quality-adjusted progression free survival (QAPFS)
* time to first subsequent treatment (TFST)
* quality-adjusted time without symptoms of toxicity (Q-TWiST)
* health related quality of life (QoL) assessed by EQ-5D-5L, FACT-ES and FACT-O questionnaires

Methods: 540 for this study eligible subjects are 1:1 allocated in this randomized, controlled, double-blinded, multi-centre study to either the test (letrozole) or control (placebo) group. The maximum maintenance treatment duration is 5 years or until symptoms of toxicity or progression of underlying disease.

Health and health-related quality of life will continuously be assessed at study entry and during routine recalls which are scheduled every 12 weeks for the first 2 years, followed by every 24 weeks for the next 3 years. Procedures performed to assess the participants' health are the same as are performed during the regular routine ovarian cancer follow-up visits: blood tests, physical as well as gynaecological examinations and may include imaging. In addition, the participants are asked to complete during the study quality of life (QoL) specific questionnaires and wear an activity tracker for one week just before the scheduled visits. These assessments will be used for the evaluation of letrozole's efficacy and burden in comparison to the standard maintenance treatment. Survival follow-up data after the mainentance treatment duration of 5 years (study end) are obtained for up to another 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Willing and able to attend the visits and to understand all study-related procedures.
* Primary, newly diagnosed FIGO Stage II to IV and histologically confirmed low or high grade serous or endometrioid epithelial ovarian/fallopian tube/peritoneal cancer
* (Interval-) debulking performed ECOG-Performance Status 0-2
* Signed informed consents (ICF-1; ICF-2)
* Paraffin-embedded tissue or paraffin-embedded cell block (from ascites) available
* Positivity (≥ 1%) for ER expression (only determined by Histopathology Core Facility of MATAO trial)
* At least 4 cycles of platinum-based chemotherapy (neoadjuvant allowed)
* Negative serum pregnancy test in women of childbearing potential who will get/have gotten a surgical resection or radiation sterilization, prior to the intervention in the therapeutical maintenance setting.

Exclusion Criteria:

* Progressive disease at the end of adjuvant treatment as defined in chapter 9.2.1 of protocol
* Women of childbearing potential (not having undergone a surgical or radiation sterilization and not getting a surgical resection, prior to the intervention in the therapeutical maintenance setting)
* Pregnant or lactating women
* Any other malignancy within the last 5 years which has impact on the prognosis of the patient
* < 4 cycles of chemotherapy in total
* Contraindications to endocrine therapy
* Inability or unwillingness to swallow tablets
* Patients with a known intolerance to galactose, lactase deficiency and glucose-galactose malabsorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 540 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) for each study group | Up to approximately 12 years
  PFS defined as the time from the date of first IMP administration until the date of progression (recurrence) or death by any cause in the absence of progression.
  Assessment of progression (recurrence) is generally indicated by SYMPTOMS and will be assessed by the investigator most commonly on the basis of CT scans of the pelvis, abdomen and thorax, according to RECIST v1.1 criteria recommended and mostly presented by an elevated CA-125 level. Elevated CA-125 levels alone shouldn't be considered as progression. Progression assessment according to local standard of care, however, is similarly acceptable.

SECONDARY OUTCOMES:
Overall survival (OS) for each study group | Up to approximately 12 years
  OS defined for each patient as the time from the date of first IMP administration until the date of death from any cause. Patients not having an event at the time of analysis will be censored at the date they were last known to be alive.
Quality-adjusted progression free survival (QAPFS) for each study group | Up to approximately 12 years
  QAPFS defined as the time from the date of first IMP administration until the date of progression (recurrence) or death by any cause in the absence of progression under consideration of the quality of life during this period. QAPFS incorporates progression-free survival (quantity) and quality of life during this period into a measure of net clinical benefit:
  QAPFS = PFS (years or months) x QoL (utility value).
  Utility values derived from the EQ-5D-L5 questionnaire will be used.
Time to first subsequent treatment (TFST) for each study group | Up to approximately 12 years
  TFST defined for each patient as the time from the date of first IMP administration until the date the patient started the next (second-line) subsequent anticancer treatment. Patients not receiving a subsequent anticancer treatment at the time of analysis will be censored at the date they were last known to be alive.
Quality-adjusted time without symptoms of toxicity (Q-TWiST) for each study group | Up to approximately 12 years
  Q-TWiST defined as the Quality adjusted Time Without appearance of any Symptoms of Toxicity related to either the progression of the cancer or side effects of the trial medication from the date of first IMP administration until dead.
  The Q-TWiST analysis considers the following three health states:
  * (1) the period experiencing toxicity (TOX)
  * (2) the period before progression without experiencing toxicity (TWiST)
  * (3) the period after relapse (REL)
  These periods are assigned preference utilities (u), which will be derived using the generic EQ-5D-5L questionnaire.
  The Q-TWiST will be calculated as the weighted sum of the time spent in each health state:
  Q-TWiST = uTox*TOX + TWiST + uRel*REL where u denotes the assigned utility for each respective health state.
Health related quality of life (QoL) assessed byFunctional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire for each study group | Up to approximately 5.25 years
  Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) is included into the study to more specifically assess the side effects from the IMPs on quality of life. The minimum value is 0, the maximum value for the specific 19 item Endocrine Symptom Subscale (ESS-19) is 76. The higher the score, the better the QOL
Health related quality of life (QoL) assessed by Functional Assessment of Cancer Therapy - Ovarian (FACT-O) questionnaire for each study group | Up to approximately 5.25 years
  In the context of this study the specific ovarian cancer symptom-oriented questionnaire Functional Assessment of Cancer Therapy - Ovarian (FACT-O) is included to assess the progression/recurrence of ovarian cancer on Quality of Life. The minimum value is 0, the maximum value including the specific Ovarian Cancer Subscale (OCS) is 152. The higher the score, the better the QOL

CONTACTS AND LOCATIONS:
Overall Officials: Heinzelmann-Schwarz, Prof. MD PhD, Principal Investigator — University Hospital Basel, Head Women's Hospital
Locations (53):
- Austria (8):
  - Krankenhaus der Barmherzigen Brüder Graz, Graz
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Landeskrankenhaus Hochsteiermark Leoben, Leoben
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Universitätsklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
  - Klinik Hietzing Wien, Vienna
- Germany (23):
  - Charité - Universitätsmedizin Berlin Campus Virchow Klinikum, Berlin
  - St. Elisabeth-Krankenhaus, Cologne
  - Donauisar Klinikum, Deggendorf
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Evangelische Kliniken Essen Mitte GmbH, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - University Hospital Freiburg, Freiburg im Breisgau
  - The University Medical Center Hamburg-Eppendorf, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Hamburg
  - Gynäkologisch-Onkologische Gemeinschaftspraxis Dres. med. C.Uleer/J.Y.Pourfard, Hildesheim
  - Klinikum Konstanz, Konstanz
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - University Hospital Münster, Münster
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - SL Klinikum Rosenheim, Rosenheim
  - Leopoldina Krankenhaus der Stadt Schweinfurt, Schweinfurt
  - Universitätsklinik Ulm, Ulm
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - AMO Wolfsburg / AMO MVZ GmbH, Wolfsburg
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Switzerland (22):
  - Kantonsspital Aarau AG, Aarau, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Oncology Institute of Southern Switzerland (IOSI)-Ente Ospedaliero Cantonale (EOC), Bellinzona, Canton Ticino
  - Centre Hospitalier du Valais Romand, Sion, Valais
  - Kantonsspital Baden AG, Baden
  - Basel Claraspital AG, Basel
  - Universitätsklinik für Medizinische Onkologie, Inselspital, Bern
  - Praxis im Frauenzentrum Lindenhofspital, Bern
  - Kantonspital Graubünden (KSGR),, Chur
  - Kantonsspital Frauenfeld, Frauenfeld
  - Hôpitaux Universitaires de Genève, Geneva
  - Frauenklinik Spital Grabs, Grabs
  - Universitätsspital Waadt/ CHUV, Lausanne
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Tumorzentrum Hirslanden Klinik St. Anna, Lucerne
  - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Klinik für Onkologie und Hämatologie Hirslanden Zürich AG, Zurich
  - Stadtspital Triemli, Zurich
  - Unispital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLaughlin PMJ, Klar M, Zwimpfer TA, Dutilh G, Vetter M, Marth C, du Bois A, Schade-Brittinger C, Reuss A, Bommer C, Kurzeder C, Heinzelmann-Schwarz V. Maintenance Therapy with Aromatase Inhibitor in epithelial Ovarian Cancer (MATAO): study protocol of a randomized double-blinded placebo-controlled multi-center phase III Trial. BMC Cancer. 2022 May 6;22(1):508. doi: 10.1186/s12885-022-09555-8. PMID 35524184